CLINICAL TRIAL: NCT05668819
Title: Open-Label, Randomized, Controlled, Parallel Group Study Evaluating Efficacy and Safety of Digital Therapeutic (TH-001) for the Treatment of Prediabetes in Adults
Brief Title: Efficacy and Safety of Digital Therapeutic in Adults With Prediabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tesu Saglik Teknolojileri A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TH001_1001
Record Dates: First submitted 2022-12-17; First posted 2022-12-30 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: PreDiabetes
Keywords: Prediabetic State; Digital Therapeutic; Mobile Health; Digital Health; Mobile Apps; Lifestyle Modification; mHealth
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized, Controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TH-001 (Experimental)
  Interventions: Device: TH-001
- Control (No Intervention)

INTERVENTIONS:
Device: TH-001 — TH001 is a software program intended to treat adults with prediabetes.
  Arms: TH-001

SUMMARY:
The study aims to evaluate the efficacy and safety of a digital therapeutic (TH-001) for adult individuals with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with prediabetes according to the ADA Prediabetes Diagnostic Criteria (the presence of at least one of the following criteria is sufficient for diagnosis: FBG 100 - 125 mg/dL, OGTT 2 hour BG: 140 - 199 mg/dL, HbA1c: 5.7% - 6.4)
* Not using medication for the treatment of prediabetes, and if so, taking a break for at least two weeks
* Having a smartphone with an iOS or Android operating system
* Being able to use a mobile application

Exclusion Criteria:

* Being diagnosed with diabetes mellitus
* Having a disease that can cause prediabetes
* Taking medication that may cause prediabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 90 days
  The difference in the mean change from baseline in HbA1c (%) at Day 90 between groups.
Change in FPG | 90 days
  The difference in the mean change from baseline in FPG (mg/dL) at Day 90 between groups.
Change in PPG | 90 days
  The difference in the mean change from baseline in 2-hour 75 g OGTT (mg/dL) at Day 90 between groups.

SECONDARY OUTCOMES:
Change in weight | 90 days
  The difference in the mean change from baseline in weight (kg) at Day 90 between groups.
Change in BMI | 90 days
  The difference in the mean change from baseline in BMI (kg/m^2) at Day 90 between groups.
Change in WC | 90 days
  The difference in the mean change from baseline in Waist Circumference (centimeters) at Day 90 between groups.
Change in WHR | 90 days
  The difference in the mean change from baseline in waist-to-hip ratio (WHR) (waist circumference and hip circumference measured in centimeters) at Day 90 between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Cakmak, MD, Principal Investigator — Istinye University Health Practice and Research Center Gaziosmanpasa Hospital
Locations (1):
- Istinye University Health Practice and Research Center Gaziosmanpasa Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cakmak R, Tosun I, Avcu H, Birer GC, Akgul O, Saini KS, Carnell J, Kutlu O. A randomised clinical trial to evaluate a digital therapeutic (TH-001) for improving glycaemic control in adults with prediabetes. Digit Health. 2025 Sep 12;11:20552076251376260. doi: 10.1177/20552076251376260. eCollection 2025 Jan-Dec. PMID 40949672